CLINICAL TRIAL: NCT05621317
Title: A Safety and Efficacy Study of PVX108 in Children and Adolescents With Peanut Allergy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aravax Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVX-201
Record Dates: First submitted 2022-10-27; First posted 2022-11-18 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Peanut Allergy; Peanut Hypersensitivity; Peanut-Induced Anaphylaxis; Immune System Diseases
Keywords: Peanut allergy; Arachis; Child; Adolescent; Immunotherapy
MeSH Terms: conditions — Peanut Hypersensitivity; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- PVX108 50 nmol in adolescents (Experimental): Twelve 4-weekly intradermal (ID) doses of PVX108 at 50 nmol in adolescents (Cohort 1)
  Interventions: Biological: PVX-108
- Placebo in adolescents (Placebo Comparator): Twelve 4-weekly ID doses of placebo matching PVX108 in adolescents (Cohort 1)
  Interventions: Biological: Placebo
- PVX108 5 nmol in children (Experimental): Twelve 4-weekly ID doses of PVX108 at 5 nmol in children (Cohort 2)
  Interventions: Biological: PVX-108
- PVX108 50 nmol in children (Experimental): Twelve 4-weekly ID doses of PVX108 at 50 nmol in children (Cohort 2)
  Interventions: Biological: PVX-108
- Placebo in children (Placebo Comparator): Twelve 4-weekly ID doses of placebo matching PVX-108 in children (Cohort 2)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PVX-108 — PVX108 comprises a mixture of peptides that represent sequences from peanut allergens
  Arms: PVX108 5 nmol in children; PVX108 50 nmol in adolescents; PVX108 50 nmol in children
Biological: Placebo — Matching placebo comprises the formulation vehicle without peptides
  Arms: Placebo in adolescents; Placebo in children

SUMMARY:
The overall aims of this study are to demonstrate that treatment with PVX108 immunotherapy has an acceptable safety profile and is effective for reducing clinical reactivity to peanut protein in children and adolescents with peanut allergy.

ELIGIBILITY:
Key Inclusion Criteria:

* Physician-diagnosed immunoglobulin E (IgE) mediated peanut allergy;
* Peanut specific serum IgE measured by ImmunoCAP® ≥ 0.7 kilounit allergy specific antibody per litre (kUA/L) at screening;
* Positive skin prick test to peanut with mean wheal diameter ≥5 mm greater than negative control at screening;
* Positive peanut double blind placebo-controlled food challenge (DBPCFC) with a reactive dose ≤300 mg peanut protein (≤443 mg cumulative reactive dose [CRD]);
* Able to perform spirometry or peak expiratory flow. Children who are 4 years of age at Screening Stage 1 visit and unable to perform peak expiratory may be enrolled providing they had no clinical features of moderate or severe persistent asthma within 1 year prior to the Screening visit;
* Forced expiratory volume in 1 second (FEV1) ≥80% predicted in adolescents and children with asthma capable of performing spirometry, or peak expiratory flow ≥80% predicted in participants with asthma unable to perform spirometry (at investigator's discretion).

Key Exclusion Criteria:

* History of or current clinically significant medical conditions or laboratory abnormalities which in the opinion of the investigator would jeopardise the safety of the participant or the validity of the study results;
* Severe or unstable asthma as assessed by the Global Initiative for Asthma (GINA) assessment of asthma control OR current treatment for asthma at GINA ≥Step 4 level;
* Participants with skin disorders that would hinder skin prick testing and/or its interpretation or study drug administration (eg, severe generalised poorly controllable atopic dermatitis);
* Any medical condition in which epinephrine (adrenaline) is contraindicated;
* Prior therapy aimed at desensitising peanut allergy, either in a formal study or in clinical practice;
* Severe or life-threatening reaction during the screening food challenge, at investigator discretion.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Ratio of maximum tolerated dose (MTD) of peanut protein at the Week 46 double blind placebo-controlled food challenge (DBPCFC) relative to baseline in children aged 4 to 11 years treated with PVX108 compared to placebo | 46 weeks

SECONDARY OUTCOMES:
Ratio of MTD of peanut protein at the Week 71 DBPCFC relative to baseline in children aged 4 to 11 years treated with PVX108 compared to placebo | 71 weeks
Percentage of children aged 4 to 11 years treated with PVX108 who achieve an MTD of at least 300 mg, 600 mg and 1000 mg at the Week 46 DBPCFC compared to placebo | 46 weeks
Percentage of children aged 4 to 11 years treated with PVX108 who achieve an MTD of at least 300 mg, 600 mg and 1000 mg at the Week 71 DBPCFC compared to placebo | 71 weeks
Ratio of cumulative reactive dose (CRD) of peanut protein at the Week 46 DBPCFC relative to baseline in children aged 4 to 11 years treated with PVX108 compared to placebo | 46 weeks
Ratio of CRD of peanut protein at the Week 71 DBPCFC relative to baseline in children aged 4 to 11 years treated with PVX108 compared to placebo | 71 weeks
Percentage of treatment responders at the Week 46 DBPCFC in children aged 4 to 11 years treated with PVX108 compared to placebo | 46 weeks
Percentage of treatment responders at the Week 71 DBPCFC in children aged 4 to 11 years treated with PVX108 compared to placebo | 71 weeks
Frequency of events of each severity grade during the Week 46 DBPCFC in children aged 4 to 11 years treated with PVX108 compared to placebo | 46 weeks
Frequency of events of each severity grade during the Week 71 DBPCFC in children aged 4 to 11 years treated with PVX108 compared to placebo | 71 weeks
Treatment emergent adverse events (TEAEs) and Serious adverse events (SAEs) during 45 weeks treatment and 26 weeks following treatment with PVX108 compared to placebo | Up to 74 weeks
  Incidence and severity of TEAEs (graded according to FDA Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers, 2007) including SAEs, TEAEs leading to study discontinuation, anaphylaxis with temporal association to investigational product (IP) administration, use of epinephrine (adrenaline) as rescue medication after IP administration, and injection site reactions.
Change from baseline in peak expiratory flow | Up to 73 weeks
Severity of symptoms upon unintentional exposure to peanut (graded according to FDA Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers, 2007) | Up to 73 weeks
Incidence of anti-drug antibodies (ADAs) associated with clinically significant TEAEs | Up to 46 weeks
Number of participants with abnormal physical examination data | Up to 74 weeks
Incidence of concomitant medication use | Up to 74 weeks
Number of participants with abnormal clinical laboratory data | Up to 74 weeks
Number of participants with abnormal vital signs | Up to 74 weeks

OTHER OUTCOMES:
Ratio of MTD of peanut protein at the Week 46 DBPCFC relative to baseline in adolescents aged 12 to 17 years treated with PVX108 compared to placebo | 46 weeks
Ratio of MTD of peanut protein at the Week 71 DBPCFC relative to baseline in adolescents aged 12 to 17 years treated with PVX108 compared to placebo | 71 weeks
Percentage of adolescents aged 12 to 17 years treated with PVX108 who achieve an MTD of at least 300 mg, 600 mg and 1000 mg at the Week 46 DBPCFC compared to placebo | 46 weeks
Percentage of adolescents aged 12 to 17 years treated with PVX108 who achieve an MTD of at least 300 mg, 600 mg and 1000 mg at the Week 71 DBPCFC compared to placebo | 71 weeks
Ratio of CRD of peanut protein at Week 46 DBPCFC relative to baseline in adolescents aged 12 to 17 years treated with PVX108 compared to placebo | 46 weeks
Ratio of CRD of peanut protein at Week 71 DBPCFC relative to baseline in adolescents aged 12 to 17 years treated with PVX108 compared to placebo | 71 weeks
Percentage of treatment responders at the Week 46 DBPCFC in adolescents aged 12 to 17 years treated with PVX108 compared to placebo | 46 weeks
Percentage of treatment responders at the Week 71 DBPCFC in adolescents aged 12 to 17 years treated with PVX108 compared to placebo | 71 weeks
Frequency of events of each severity grade during the Week 46 DBPCFC in adolescents aged 12 to 17 years treated with PVX108 compared to placebo | 46 weeks
Frequency of events of each severity grade during the Week 71 DBPCFC in adolescents aged 12 to 17 years treated with PVX108 compared to placebo | 71 weeks
Changes from baseline in allergen specific immunoglobulins after 45 weeks treatment with PVX108 compared to placebo | Up to 74 weeks
Changes from baseline in cellular immune response after 45 weeks treatment with PVX108 compared to placebo: Exploratory | Up to 74 weeks
Changes from baseline in titrated peanut skin prick test (SPT) response after 45 weeks treatment with PVX108 compared to placebo | Up to 74 weeks
Proportion of participants in each cohort who develop treatment-induced or treatment-enhanced ADAs during 45 weeks treatment with PVX108 compared to placebo | 45 weeks
Change from baseline in Food Allergy Related Quality of Life Questionnaire Child Form (FAQLQ-CF) score (Range 1-7, higher score indicates worse outcome) at Week 46 and at Week 71 in children enrolled in Cohort 2 treated with PVX108 compared to placebo | Up to 71 weeks
Change from baseline in FAQLQ-Teenager Form (FAQLQ-TF) score (Range 1-7, higher score indicates worse outcome) at Week 46 and at Week 71 in adolescents enrolled in Cohort 1 treated with PVX108 compared to placebo | Up to 71 weeks
Change from baseline in Food Allergy Independent Measure (FAIM) score (Range 1-7, higher score indicates worse outcome) at Week 46 and at Week 71 in children enrolled in Cohort 2 treated with PVX108 compared to placebo | Up to 71 weeks
Change from baseline in FAIM score (Range 1-7, higher score indicates worse outcome) at Week 46 and at Week 71 in adolescents enrolled in Cohort 1 treated with PVX108 compared to placebo | Up to 71 weeks
Change from baseline in FAQLQ-Parent Form (FAQLP-PF) score (Range 1-7, higher score indicates worse outcome) at Week 46 and at Week 71 in children enrolled in Cohort 2 treated with PVX108 compared to placebo | Up to 71 weeks
Change from baseline in FAQLQ-Parent Form Teenager (FAQLQ-PFT) score (Range 1-7, higher score indicates worse outcome) at Week 46 and at Week 71 in adolescents enrolled in Cohort 1 treated with PVX108 compared to placebo | Up to 71 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian Vickery, MD, Principal Investigator — Emory University
Locations (14):
- United States (8):
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Riley Children's Hospital at IU, Indianapolis, Indiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - IAA Clinical Research, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Australia (6):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Women's and Children's Hospital, North Adelaide, South Australia
  - The Royal Children's Hospital Melbourne, Parkville, Victoria
  - Perth Children's Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No